CLINICAL TRIAL: NCT06631664
Title: Contribution of Reciprocal Electrical Stimulation Across Elbow Muscles in Motor Recovery of Infants With Erbs Palsy: a Randomized Controlled Trial
Brief Title: Electrical Stimulation on Erbs Palsy Infants
Acronym: RES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Collaborators: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Hend Reda Sakr, Lecturer of Physical Therapy, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hend 6
Record Dates: First submitted 2024-09-29; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Erbs Palsy
Keywords: Brachial plexus birth injury; Neuromuscular electrical stimulation; Active motion; Electroneurography; Motor function
MeSH Terms: conditions — Brachial Plexus Neuropathies

STUDY DESIGN:
Intervention Model Description: A prospective single-blind randomized clinical trial
Who Masked: Investigator
Masking Description: The investigator was blinded to the interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study group (Experimental): Twenty children suffering from Obstetric brachial plexus injury limited to nerve roots C5, C6, with/without involvement of C7
  Interventions: Other: Traditional physical therapy; Device: A computerized electrical stimulator (Vectra®2C; Chattanooga, TS, USA)
- Control group (Other): Twenty children suffering from Obstetric brachial plexus injury limited to nerve roots C5, C6, with/without involvement of C7
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Other: Traditional physical therapy — Participants received a traditional physical therapy program three times a week, for three successive months. Each session lasted for approximately 30 minutes and composed of the following: 1) Massage (spiral effleurage, longitudinal and transverse thumb effleurage for 5 minutes or until hyperemia), 2) Facilitation of muscle contraction through a variety of tactile and proprioceptive stimulation techniques - this was applied for the shoulder flexors, abductors, and external rotators, elbow flexors, and wrist/finger extensors. In patients whose lesion extend to involve C7, The facilitation techniques were also applied to elbow extensors. 3) Weight-bearing exercise, considering the developmental milestone (prone forearm support, prone full hand support). 4) Range of motion exercises - all joints of the affected side were moved through the full range of motion. 5) Sucking exercise.
Device: A computerized electrical stimulator (Vectra®2C; Chattanooga, TS, USA) — The patient was positioned in supine lying position with the affected arm beside the body and elbow extended, the skin over the anterior and posterior comportment of the upper arm was cleaned using medical cotton sacked in alcohol before the application.
  The first two stimulating electrodes for the biceps muscle were placed at the superior and inferior 1/3 of anterior surface of the upper arm with a distance in between the two electrodes at least the size of one of them, while the other two electrodes for the triceps muscle were placed at the superior and inferior 1/3 of the posterior surface of the upper arm.
  One millisecond pulse duration and a frequency of 50Hz with a rectangular shaped pulse were utilized and stimulation was applied for 15 minutes. At first a low-intensity current is applied and gradually increased till a gentle contraction of the muscles appears and allow time for the child to become accustomed to the current and maintained sufficient and observable contraction.
  Arms: Study group

SUMMARY:
This study examined the effect of reciprocal electrical stimulation (RES) across elbow flexors and extensors on the reaction of degeneration percentage and motor function in Erbs palsy infants.

Forty infants with Erb's palsy aged between 2-5 months were randomly allocated to one of two equal groups: the control group (A) received standard physical therapy, the study group (B) received traditional physical therapy plus a 15-minute RES through elbow flexors and extensors. For three months, interventions were carried out three times each week. The percentage of degeneration and motor function reaction were assessed pre-and post-treatment using electromyography and Toronto active motion scale, respectively.

DETAILED DESCRIPTION:
This study examined the effect of reciprocal electrical stimulation (RES) across elbow flexors and extensors on the reaction of degeneration percentage and motor function in Erbs palsy infants.

Forty infants with Erb's palsy aged between 2-5 months were randomly allocated to one of two equal groups: the control group (A) received standard physical therapy, the study group (B) received traditional physical therapy plus a 15-minute RES through elbow flexors and extensors. For three months, interventions were carried out three times each week. The percentage of reaction of degeneration and motor function were assessed pre-and post-treatment using electromyography and the Toronto active motion scale respectively.

ELIGIBILITY:
Inclusion Criteria:

* Infants with OBPI limited to nerve roots C5, C6, with/without involvement of C7, partial lesion as determined by electrophysiological examinations, age between two to five months, and willingness of the infant's family to take part in the study.

Exclusion Criteria:

* Infants with clavicular or humeral fractures, complete transection of nerve roots, other neurological co-morbidities such cerebral palsy, congenital musculoskeletal deformities, or recommendation against electrical stimulation by the attending neuro-pediatrician.

Ages: 2 Months to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-04-23 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
Percentage of degeneration | 2 months
  Surface electrodes were used in a computerized electromyographic device (Neuro screen plus four channel-version, TOENNES 97204 Hochberg, Germany) to calculate the percentage of degeneration of the biceps and triceps brachii muscles.
  A 1 Hz frequency and 5 ms time basis were used to create a rectangular pulse. The strength of the stimulating current was gradually raised until there was no further rise in the amplitude of the diphasic myogenic compound action potential. A 10% increase in current was given to assure supramaximal stimulation. The level of stimulation ranges from 15 to 40 mA. The Neuro screen plus system's software was used to calculate the peak-to-peak amplitude. The following equation was used to compute the percentages of degeneration:
  RD= 100{Amplitude of evoked response(in µv) affected side/Amplitude of evoked response(in µv)normal side x 100}
Toronto active motion scale (TAMS) | 2 months
  The motor recovery was assessed using the Toronto Active Motion Scale (TAMS). For this study, scores for elbow flexion and extension were recorded.
  It consists of 15 movements of upper limb joints with an eight-point scale measuring the strength of these movements, first by measuring the range of motion at each joint with gravity eliminated, and then measuring the range of motion against gravity. The scoring of the TAMS is defined as follows:
  Observation Gravity elimination Muscle grade
  No muscle contraction 0 Contraction, no movement 1 Motion < range 2 Motion > range 3 Full range of movement 4
  Against gravity Motion < range 5 Motion > range 6 Full range of movement 7

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sattam bin Abdul-Aziz University, Al Kharj, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No